CLINICAL TRIAL: NCT01289249
Title: Meropenem Plasma Concentration Measurements at the Pediatric Medical Ward, Oslo University Hospital, Rikshospitalet
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2010/3023-1
Record Dates: First submitted 2011-01-31; First posted 2011-02-03 (Estimated); Last update posted 2014-11-06 (Estimated); Status verified 2014-11

CONDITIONS: Bacterial Infection
Keywords: meropenem; child; bacterial infection; treatment evaluation
MeSH Terms: conditions — Bacterial Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Two blood samples are taken from each included patient. (Each 2 ml heparin full blood).
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Children receiving meropenem: Children aged from 3 months to 18 years that receive treatment with meropenem.

SUMMARY:
The object of the study is to investigate whether all included patients receive treatment that is effective against all bacteria that are defined as sensitive to meropenem with the current treatment regimen. Will the investigators findings motivate routine monitoring of plasma concentrations in children receiving meropenem? Up to 50 patients will be included in the study, and all participants are children.

ELIGIBILITY:
Inclusion Criteria:

* Children aged from 3 months to 18 years that receive treatment with meropenem. Inclusion is independent of how long the patient has been receiving treatment. Children receiving other treatment (except hemodialysis)/other medications can be included.

Exclusion Criteria:

* Children less than three months of age. Patients receiving hemodialysis. Lack of consent.

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients at the Pediatric medical ward.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2011-01; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
We will determine how many of the patients in our material that have plasma concentrations of meropenem above 8 mg/l for at least 40% and 75% of the time. | 1 dosing interval (8 hours)

CONTACTS AND LOCATIONS:
Overall Officials: Odd Brørs, Dr Med, Study Director — Oslo University Hospital; Margrete L Burns, BMed, Study Chair — Oslo univeristy hospital; Øystein Riise, PhD, Study Chair — Oslo University Hospital; Tore Abrahamsen, Dr Med, Study Chair — Oslo univeristy hospital; Gaut Gadeholt, Dr Med, Study Chair — Oslo University Hospital
Locations (1):
- Oslo univeristy hospital, Rikshospitalet, Oslo, Norway

REFERENCES:
- [Background] Ikeda K, Ikawa K, Morikawa N, Miki M, Nishimura S, Kobayashi M. High-performance liquid chromatography with ultraviolet detection for real-time therapeutic drug monitoring of meropenem in plasma. J Chromatogr B Analyt Technol Biomed Life Sci. 2007 Sep 1;856(1-2):371-5. doi: 10.1016/j.jchromb.2007.05.043. Epub 2007 Jun 6. PMID 17581801